CLINICAL TRIAL: NCT01862289
Title: Prevalence of Hyperventilation Syndrome in Difficult Asthmatics Uncontrolled Despite a Daily Maximal Doses of Inhaled Treatment
Brief Title: Prevalence of Hyperventilation Syndrome in Difficult Asthma
Acronym: PRESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P110904; CRC 11093 (Other: APHP - Clinical research department)
Record Dates: First submitted 2013-05-22; First posted 2013-05-24 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Difficult Asthma; Severe Persistent Asthma; Hyperventilation Syndrome
Keywords: difficult asthma; hyperventilation syndrome; prevalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe uncontrolled asthma (Experimental): Asthmatics patients with uncontrolled symptoms despite a daily treatment by high doses of inhaled steroids and LABA. Diagnostic of chronic hyperventilation syndrome.
  Interventions: Other: Diagnostic of chronic hyperventilation syndrome

INTERVENTIONS:
Other: Diagnostic of chronic hyperventilation syndrome — Nijmegen questionnaire, Hyperventilation challenge and blood gases
  Other Names: Exploration to sarch a chronic hyperventilation syndrome

SUMMARY:
Most of asthmatics patients remain uncontrolled despite an inhaled steroids treatment. Chronic hyperventilation syndrome (also called Idiopathic Hyperventilation) occurs in 20 to 40% of asthmatic patients. The purpose of the study is to assess the prevalence of chronic hyperventilation syndrome in a specific population of difficult-to-treat asthmatics patients, those who receive daily high doses of inhaled steroids (≥ 1000 µg of fluticasone with an additional treatment by a long-acting beta 2-agonist (LABA) and who remain uncontrolled (Asthma control test (ACT) < 18). We plan to realize a systematic assessment of the diagnosis of chronic hyperventilation syndrome with the Nijmegen questionnaire, blood gases at rest, hyperventilation testing and Cardiopulmonary Exercise Testing(CPET). We also will collect demographic information as well as information about asthma history, asthma control and treatment.

DETAILED DESCRIPTION:
There is only one visit. During this visit, each patient will complete self-questionnaires like Nijmegen, Hospital Anxiety and Depression Scale(HAD), Short-Form 36(SF36), and Asthma Quality of Life Questionnaire (AQLQ), The participants will have baseline spirometry and fractional exhaled nitric oxide measured at expiratory flow of 50 mL/s (FENO50), blood gases at rest, an hyperventilation challenge and Cardiopulmonary Exercise Testing(CPET) to determine accurately the presence or not of chronic hyperventilation syndrome. The diagnosis is confirmed by two positive tests (Nijmegen, Hyperventilation challenge and blood gases) and the final decision of a medical committee. The first step is to determine the prevalence oh this syndrome in this specific population. The second step is to assess the sensitivity, the specificity, the false positive rate and the false negative rate of the different parameters measured during the tests.

ELIGIBILITY:
Inclusion Criteria:

* men and women,
* aged more than 18,
* non smokers for two years or longer, less than 10 pack/years smoking history,
* physician-diagnosed asthma,
* uncontrolled asthma with Asthma control test (ACT) < 18,
* historical of FEV1 reversibility,
* daily inhaled steroids treatment by at least 2000microg eq beclomethasone,
* Forced expiratory volume in 1 second (FEV1) > 50% predicted value

Exclusion Criteria:

* other chronic pulmonary disease,
* vocal cord dysfunction,
* pregnancy,
* Participation in another interventional research trial,
* unable to provide consent,
* asthma exacerbation within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-04-28 (Actual); Primary Completion 2016-10-18 (Actual); Study Completion 2016-10-18 (Actual)

PRIMARY OUTCOMES:
Diagnostic of the hyperventilation syndrome | Up to 4 hours
  value of Nijmegen questionnaire, of blood gases at rest, of hyperventilation testing and of CPET

SECONDARY OUTCOMES:
Assess the diagnosis value of the nijmegen questionnaire. | Up to 4 hours
Assess the diagnosis value of the blod gases at rest. | up to 4 hours
Assess the diagnosis value of the hyperventilation challenge. | Up to 4 hours
Assess the diagnosis value of the CPET. | Up to 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Garcia, MD, PhD, Principal Investigator — Assistance Publique Hôpitaux de Paris - Bicêtre Hospital
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Bicêtre Hospital, Le Kremlin-Bicêtre, France